CLINICAL TRIAL: NCT05426980
Title: Artificial Intelligence in Predicting Progression in Multiple Sclerosis Study
Acronym: AI ProMiS
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Collaborators: Novartis (Industry); General and Teaching Hospital Celje (Other); University Medical Centre Ljubljana (Other); University Medical Centre Maribor (Other); Izola General Hospital (Other)
Responsible Party: Principal Investigator, Ziga Spiclin, Associate professor, PhD, University of Ljubljana
Other Study IDs: 0120-570/2021/5
Record Dates: First submitted 2022-05-26; First posted 2022-06-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis Lesion; Multiple Sclerosis Brain Lesion
Keywords: Artificial intelligence; Prediction model; Magnetic resonance imaging; Computer-assisted image analysis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study proposal focuses on multiple sclerosis (MS), a chronic incurable disease of the central nervous system (CNS). The MS disease is characterised by recurrent transient disability progression, quantified by increase in the extended disability status score (EDSS), and subsequent remission (disappearance of symptoms and reduced EDSS score) or, alternatively, a gradual EDSS disability progression and exacerbation of associated symptoms. At the same time, the MS is characterised by multifocal inflammatory lesions disseminated throughout the white and grey matter of the CNS, which can be observed and quantified in the magnetic resonance (MR) scans. The proposed study will address the critical unmet need of computer-assisted extraction and assessment of prognostic factors based from an individual patient's brain MR scan, such as lesion count, volume, whole-brain and regional brain atrophy, and atrophied lesion volume, in order to evaluate the capability for personalized future disability progression prediction.

ELIGIBILITY:
Inclusion Criteria:

* persons diagnosed with MS (any phenotype; according to the 2010 McDonald criteria) and CIS patients
* availability of at least two MRI exams with both FLAIR and T1-weighted scans of the same participant over a period of at least 6 months at the most recent examination
* availability of demographic, clinical data and treatment information for the same participant over a period of at least 6 months at the most recent examination
* availability of EDSS score and at least one previous EDSS scores for the same participant over a period of at least 6 months at the most recent examination

Exclusion Criteria:

* other clinically relevant systemic diseases if the researcher considers them to be significant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be based on a retrospective secondary analysis of demographic and clinical data and MRI scans of approximately 1200 Slovenian patients with MS that are regularly monitored between 2015 and present.
Sampling Method: Non-Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Atrophied lesion volume derived from MRI predicts confirmed EDSS disability progression | Atrophied lesion volume quantified from two or more MR scans across the span of at least one and up to five years
  Patients will be divided into two groups based on the presence or absence of EDSS disability progression (DP) during the observation period. The DP converters will be classified as patients with an EDSS change of at least 1.5 if the baseline EDSS is less than 1.0, those with an EDSS change of at least 1.0 if the baseline EDSS is 1.0-5.5, and those with an EDSS change of at least 0.5 if the baseline EDSS is 5.5 or higher [15]. DP converters should have confirmed progression of EDSS impairment over a period of at least 6 months. DP non-converters include individuals who do not meet the criteria for conversion. Atrophied lesion volume will be quantified from MR scans taken >6 months prior to the observed EDSS increase. Advanced artificial intelligence based image analysis tools will be applied to assess the atrophied lesion volume.

SECONDARY OUTCOMES:
Atrophied lesion volume derived from MRI predicts conversion to secondary progressive multiple sclerosis | Atrophied lesion volume quantified from two or more MR scans across the span of least one and up to five years
  Patients will be divided into two groups, i.e. those who transitioned from clinically isolate syndrome (CIS) or relapsing-remitting (RR) to secondary progressive (SP) form of MS and those who were diagnosed with CIS/RRMS during the observation period. A consilium for patients with MS will confirm the SPMS diagnosis by consensus. Atrophied lesion volume will be quantified from MR scans taken >6 months prior to the observed conversion to the SPMS. Advanced artificial intelligence based image analysis tools will be applied to assess the atrophied lesion volume.

CONTACTS AND LOCATIONS:
Overall Officials: Ziga Spiclin, PhD, Principal Investigator — University of Ljubljana
Locations (4):
- Slovenia (4):
  - University medical center Ljubljana, Ljubljana, Osrednjeslovenska
  - General and teaching hospital Celje, Celje
  - General hospital Izola, Izola
  - University medical center Maribor, Maribor

IPD SHARING:
Plan to Share IPD: No